CLINICAL TRIAL: NCT06914986
Title: A Prospective Multicenter Randomized Controlled Trial of Flexible And Navigable Suction Ureteral Access Sheath Combined With Needle Perc for the Treatment of Partial Staghorn Renal Calculi
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24747-0-02
Record Dates: First submitted 2025-04-01; First posted 2025-04-07 (Actual); Last update posted 2025-04-07 (Actual); Status verified 2025-01

CONDITIONS: Urinary Calculi
Keywords: partial staghorn renal calculi
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Intervention Model Description: A Prospective Multicenter Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- flexible and navigable suction ureteral access sheath combined with needle perc (Experimental)
  Interventions: Procedure: Performed flexible and navigable suction ureteral access sheath combined with needle perc
- PCNL group (Other)
  Interventions: Procedure: PCNL

INTERVENTIONS:
Procedure: Performed flexible and navigable suction ureteral access sheath combined with needle perc — Patients are performed flexible and navigable suction ureteral access sheath combined with needle perc or PCNL
  Arms: flexible and navigable suction ureteral access sheath combined with needle perc
Procedure: PCNL — Patients were performed flexible and navigable suction ureteral access sheath combined with needle perc or PCNL
  Arms: PCNL group

SUMMARY:
The goal of this clinical trial is to learn if flexible and navigable suction ureteral access sheath combined with needle perc works to treat partial staghorn renal calculi. It will also learn about the safety of drug ABC. The main questions it aims to answer are:

* Does flexible and navigable suction ureteral access sheath combined with needle perc result in similar stone free rate compared with PCNL
* Does flexible and navigable suction ureteral access sheath combined with needle perc result in more complications compared with PCNL Researchers will compare flexible and navigable suction ureteral access sheath combined with needle perc result in similar stone free rate compared with PCNL to see if flexible and navigable suction ureteral access sheath combined with needle perc works to treat partial staghorn renal calculi.

Participants will:

* Performed flexible and navigable suction ureteral access sheath combined with needle perc or PCNL
* Visit the clinic after surgery 1 month and 3 month for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years
2. CT scan indicates partial staghorn calculi
3. Able to complete the study in accordance with the protocol requirements
4. Informed about the study and has signed the informed consent form

Exclusion Criteria:

1. Severe renal insufficiency (GFR < 30 ml/min/1.73 m²)
2. Significant calyceal hydronephrosis (calyceal width ≥ 2 cm)
3. Renal stone volume > 33.5 cm³
4. Renal stones or nephrocalcinosis caused by genetic diseases or definite metabolic disorders that have not been ruled out, such as renal tubular acidosis, primary hyperoxaluria, primary hyperparathyroidism, etc.
5. Congenital or structural renal abnormalities: spinal deformity, ankylosing spondylitis, horseshoe kidney, medullary sponge kidney, duplicated kidney, polycystic kidney, ectopic kidney, etc.
6. History of previous open renal stone surgery
7. Patients with uncontrolled urinary tract infections
8. Subjects deemed by the investigator to have other factors that make them unsuitable for participation in this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
stone free rate | 3 month after surgery
  Patient will have CT scan 3 month after surgery

SECONDARY OUTCOMES:
complications | 3 month after surgery
  Patients were recorded complications after surgery

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code